CLINICAL TRIAL: NCT04351932
Title: Bone Marrow Versus Adipose Autologous Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis: A Randomized Non Blind Controlled Clinical Trial
Brief Title: Bone Marrow Versus Adipose Autologous Mesenchymal Stem Cells for the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Catolica Santiago de Guayaquil (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Carlos Chiriboga Accini, Research Professor. Orthopaedic Staff. Omnihospital., Universidad Catolica Santiago de Guayaquil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSantiagodeGuayaquil001
Record Dates: First submitted 2019-05-04; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Osteo Arthritis Knee
Keywords: Mesenchymal stem cell

STUDY DESIGN:
Intervention Model Description: A total of 54 patients with the diagnosis of knee OA grade II and III will be recruited to receive a single intra-articular injection of MSC: Group 1 (n 18 patients) will receive BM-MSC, Group 2 (n 18 patients) will receive AD-MSC. Group 3 (18 patients) will receive a combination of BM-MSC and AD-MSC.
Masking Description: A randomized non blind clinical trial with active control. For this purpose, the random number generator, found on the RANDOM.ORG ® website (available at https://www.random.org/integers/)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bone marrow mesenchymal stem cell (Active Comparator): Bone marrow mesenchymal stem cells 10 cc by intra articular injection once
  Interventions: Biological: bone marrow mesenchymal stem cells
- adipose mesenchymal stem cells (Active Comparator): Stromal vascular factor from adipose mesenchymal stem cells 10 cc by intra articular injection once
  Interventions: Biological: Adipose Mesenchymal stem cells
- Bone marrow and Adipose mesenchymal stem cells (Active Comparator): Bone marrow and Stromal vascular factor from adipose mesenchymal stem cells 5 cc each one, by intra articular injection once.
  Interventions: Biological: bone marrow & adipose mesenchymal stem cells injection

INTERVENTIONS:
Biological: bone marrow mesenchymal stem cells — intrarticular bone marrow mesenchymal stem cells injection
  Arms: bone marrow mesenchymal stem cell
Biological: Adipose Mesenchymal stem cells — intrarticular adipose mesenchymal stem cells injection
  Arms: adipose mesenchymal stem cells
Biological: bone marrow & adipose mesenchymal stem cells injection — intrarticular bone marrow and adipose stem cells injection.
  Arms: Bone marrow and Adipose mesenchymal stem cells

SUMMARY:
Mesenchymal stem cells (MSC) are stromal cells that have the ability to self-renew and also exhibit multilineage differentiation. MSCs can be isolated from a variety of tissues, such as umbilical cord, bone marrow, and adipose tissue. The multipotent properties of MSCs make them a promising option for the treatment of osteoarthritis (OA).

Bone marrow mesenchymal stem cells (BM-MSC) and adipose derived mesenchymal stem cells (AD-MSC) have been used separately to treat OA. The aim of the present study will be to compare in a randomized non blind controlled clinical trial 3 types of intra-articular injections containing MSC populations obtained from two clinically relevant sources: BM-MSC, AD-MSC and a combination of both BM-MSC and AD-MSC.

DETAILED DESCRIPTION:
The aim of the present study will be to compare 3 types of intra-articular injections of MSC populations obtained from two clinically relevant sources: injections containing BM-MSC or AD-MSC or a combination of both BM-MSC,and AD-MSC in a randomized non blind clinical trial.

To assess the efficacy and safety of 3 kind of MSC injections in relation to pain, function and quality of life in patients with knee OA.

A total of 54 patients with the diagnosis of knee OA grade II and III will be recruited to receive a single intra-articular injection of MSC: Group 1 (n 18 patients) will receive BM-MSC, Group 3 (n 18 patients) will receive AD-MSC. Group 3 (18 patients) will receive a combination of BM-MSC and AD-MSC.

A randomized non blind clinical trial with active control. For this purpose, the random number generator is 54, found on the RANDOM.ORG ® website (available at https://www.random.org/integers/)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years, with grade II and III knee OA, according to the Ahlbäck classification will be included.
* Minimal VAS pain score of 4.
* Chronic knee pain of mechanical origin.
* All patients who sign a specially prepared informed consent for this clinical trial.

Exclusion Criteria:

* Varus or valgus knee mal alignment superior to 10°.
* OA grade IV according Ahlbäck classification.
* Bone marrow cancer like lymphoma.
* Severe anemia.
* Active infections.
* Pregnant patients.
* Inmune diseases such as Rheumatoid arthritis, gout or pseudogout arthritis, psoriasis.
* Bone diseases such as Kahler and Paget.
* Corticoesteroid and hyaluronic injections within the last 3 months.
* Knee surgery in the last 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-06-07 (Estimated); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-09-07 (Estimated)

PRIMARY OUTCOMES:
knee pain assessed by Visual Analogue Scale. | 12 months
  psychometric response scale which used in questionnaires. It is a measurement instrument for subjective characteristics of pain . Score from O to 10. O indicate no pain, and 10 indicate the worst pain.
knee function assessed by WOMAC (Wester Ontario McMaster Osteoarthritis Index). quosteionary. | 12 months
  The Index contains 24 questions five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Individual question responses are assigned a score of between 0 (extreme) and 4 (None). Individual question scores are then summed to form a raw score ranging from 0 (worst) to 96 (best). Finally, raw scores are normalized by multiplying each score by 100/96. This produces a reported WOMAC Score of between 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Quantitative T2-Mapping Evaluation of Changes in Cartilage Matrix | 6 months after procedure
  MRI T2 mapping of the cartilage is a non-invasive functional imaging technique delivering cartography of the T2 relaxation time of the cartilage without any contrast injection. It is sensitive to tissue anisotropy, and provides compositional information on the cartilage collagen network, water content and proteoglycans concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Chiriboga, MD, Principal Investigator — Universidad Católica Santiago de Guayaquil
Locations (1):
- Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: JUNE 2021 TO SEPTEMBER 2021
Access Criteria: drcarloschiriboga@gmail.com

REFERENCES:
- [Result] Wagner W, Wein F, Seckinger A, Frankhauser M, Wirkner U, Krause U, Blake J, Schwager C, Eckstein V, Ansorge W, Ho AD. Comparative characteristics of mesenchymal stem cells from human bone marrow, adipose tissue, and umbilical cord blood. Exp Hematol. 2005 Nov;33(11):1402-16. doi: 10.1016/j.exphem.2005.07.003. PMID 16263424
- [Result] Wakitani S, Imoto K, Yamamoto T, Saito M, Murata N, Yoneda M. Human autologous culture expanded bone marrow mesenchymal cell transplantation for repair of cartilage defects in osteoarthritic knees. Osteoarthritis Cartilage. 2002 Mar;10(3):199-206. doi: 10.1053/joca.2001.0504. PMID 11869080
- [Result] Xia P, Wang X, Lin Q, Li X. Efficacy of mesenchymal stem cells injection for the management of knee osteoarthritis: a systematic review and meta-analysis. Int Orthop. 2015 Dec;39(12):2363-72. doi: 10.1007/s00264-015-2785-8. Epub 2015 May 6. PMID 25944079
- [Result] Wakitani S, Okabe T, Horibe S, Mitsuoka T, Saito M, Koyama T, Nawata M, Tensho K, Kato H, Uematsu K, Kuroda R, Kurosaka M, Yoshiya S, Hattori K, Ohgushi H. Safety of autologous bone marrow-derived mesenchymal stem cell transplantation for cartilage repair in 41 patients with 45 joints followed for up to 11 years and 5 months. J Tissue Eng Regen Med. 2011 Feb;5(2):146-50. doi: 10.1002/term.299. PMID 20603892
- [Result] Jo CH, Lee YG, Shin WH, Kim H, Chai JW, Jeong EC, Kim JE, Shim H, Shin JS, Shin IS, Ra JC, Oh S, Yoon KS. Intra-articular injection of mesenchymal stem cells for the treatment of osteoarthritis of the knee: a proof-of-concept clinical trial. Stem Cells. 2014 May;32(5):1254-66. doi: 10.1002/stem.1634. PMID 24449146
- [Result] Peeters CM, Leijs MJ, Reijman M, van Osch GJ, Bos PK. Safety of intra-articular cell-therapy with culture-expanded stem cells in humans: a systematic literature review. Osteoarthritis Cartilage. 2013 Oct;21(10):1465-73. doi: 10.1016/j.joca.2013.06.025. Epub 2013 Jul 4. PMID 23831631
- [Result] Freitag J, Bates D, Boyd R, Shah K, Barnard A, Huguenin L, Tenen A. Mesenchymal stem cell therapy in the treatment of osteoarthritis: reparative pathways, safety and efficacy - a review. BMC Musculoskelet Disord. 2016 May 26;17:230. doi: 10.1186/s12891-016-1085-9. PMID 27229856

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT04351932/Prot_SAP_000.pdf